CLINICAL TRIAL: NCT07269730
Title: Validate the Effect of T-spray on ECC in Clinical Trials
Brief Title: Validate the Effect of Calcium Oral Spray on Early Childhood Caries
Status: Completed | Type: Observational
Sponsor: Tri-Service General Hospital (Other)
Responsible Party: Principal Investigator, Da-Yo Yuh, Attending Physician, Tri-Service General Hospital
Other Study IDs: A202305084; 801GB112200 (Other Grant/Funding Number: Tri-Service General Hospital, Tapiei, Taiwan)
Record Dates: First submitted 2025-11-25; First posted 2025-12-08 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-05

CONDITIONS: Dental Caries Tooth Demineralization; Early Childhood Caries (ECC)
Keywords: ECC; Oral spray

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Biospecimen Retention: Samples With DNA — Dental biofilm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- placebo oral spray: formula 1 (0.3% calcium) oral spray
- formula 2 (0.3% calcium plus 225 ppm fluoride) oral spray
- formula 1 (0.3% calcium): Patient receiving oral spays containing 0.3% calcium solution for more than 2 month.

SUMMARY:
This study aimed to evaluate the effects of calcium-based solutions spraying on teeth to evaluate the reduction of cariogenicity through a randomized clinical trial. In the randomized clinical trial, fifteen children will be assigned to placebo, formula 1 (0.3% calcium), or formula 2 (0.3% calcium plus 225 ppm fluoride) groups of oral sprays for two months. Plaque bacterial composition, salivary calcium levels, and the cariogenicity area before and after the usage of sprays will be evaluated.

DETAILED DESCRIPTION:
Calcium has been proposed as an alternative for promoting remineralization of dental caries. This study aimed to evaluate the effects of calcium-based solutions spraying on teeth to evaluate the reduction of cariogenicity through a randomized clinical trial. In the randomized clinical trial, fifteen children will be assigned to placebo, formula 1 (0.3% calcium), or formula 2 (0.3% calcium plus 225 ppm fluoride) groups of oral sprays for two months. Plaque bacterial composition will be analyzed using 16S rRNA gene sequencing, salivary calcium levels using enzyme-linked immunosorbent assay (ELISA), and the cariogenicity area by quantitative light-induced fluorescence (QLF).

ELIGIBILITY:
Inclusion Criteria:

Required participants to have an ICDAS code ≥ 1 and ≤ 3 as determined by a clinician.

Exclusion Criteria:

1. Patient has received caries removal and restoration.
2. Patient has received fluoridation within 3 months.
3. The parents do not agree to participate in the study.
4. Patient has ICDAS code 4 - code 6

Ages: 3 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: A randomized clinical trial (RCT) will be conducted in a double-blind manner with 15 children presenting with early carious lesions in Tri-Service General Hospital, Taipei, Taiwan. Participants will be randomly assigned to one of three groups: placebo (control) and two formulations of calcium spray.
Sampling Method: Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2024-01-31 (Actual); Primary Completion 2024-08-05 (Actual); Study Completion 2025-11-11 (Actual)

PRIMARY OUTCOMES:
salivary calcium | Saliva samples will be collected at the time of recruitment and 2 months after the application of the clinical trial.
  Saliva samples collected during the clinical trial will be centrifuged at 3000 rpm for 10 minutes to obtain the clarified supernatant, which will then be diluted tenfold for calcium measurement. Calcium concentration will be determined colorimetrically using arsenazo III in an ELISA reader. The calcium-arsenazo III complex will be measured spectrophotometrically at 652 nm, with absorbance proportional to calcium concentration in the sample.

SECONDARY OUTCOMES:
Plaque bacterial composition | Plaque samples will be collected at the time of recruitment and 2 months after the application of the clinical trial.
  Three out of 15 participants will be selected for bacterial sampling (pre- and post-treatment). Plaque samples will be collected using a periodontal probe and stored in 1.5 mL tubes containing 500 μL of preservation solution at -80°C.
  Bacterial DNA will be extracted following the manufacturer's instructions using the EasyPure Bacteria Genomic DNA Kit (TransGen Biotech, Cat No. EE161). DNA purity and concentration were verified using a Nanodrop spectrophotometer. The V3 and V4 regions of the 16S rRNA gene will be amplified with primers (CCTACGGRRBGCASCAGKVRVGAAT and GGACTACNVGGGTWTCTAATCC) and the MetaVX Library Preparation Kit. Taxonomic classification will be performed using the Silva 138 reference database and the Ribosomal Database Project (RDP).

OTHER OUTCOMES:
cariogenicity area | QLF images of maxillary front teeth will be collected at the time of recruitment and 2 months after the clinical trial.
  In the clinical trial, QLF imaging produced three outputs: (1) an original photograph, (2) a binary image highlighting carious lesions, and (3) a fluorescent image. The QLF-area (%) and its change (ΔQLF-area) were measured and compared.

CONTACTS AND LOCATIONS:
Locations (1):
- Tri-Service General Hospital, Taipei, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: No
Patients who will be recruited are children under 15 years old, whose privacy should be further protected.